CLINICAL TRIAL: NCT06184919
Title: Preparing Older Adults for Major Abdominal Surgery: a Systems Engineering Approach to Implement Preoperative Comprehensive Geriatric Assessments
Brief Title: Preparing Older Adults for Major Surgery With Preoperative Comprehensive Geriatric Assessments
Status: Active, not recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2022-1516; A539707 (Other: UW Madison); SMPH/SURGERY/COLON RECT (Other: UW Madison); 1K23AG081487-01 (NIH); 2024-0044 [Aim 2] (Other: UW Madison)
Record Dates: First submitted 2023-12-13; First posted 2023-12-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Surgery; Aging; Health Care Utilization; Frailty
Keywords: Human Factors Engineering; Perioperative Optimization
MeSH Terms: conditions — Patient Acceptance of Health Care; Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients and caregivers: Patients attending the Perioperative Optimization of Senior Health (POSH) clinic
  Interventions: Other: Process Mapping: Observations; Other: Process Mapping: Interviews; Other: Participatory Design
- Healthcare providers: Healthcare providers referring to or working in the Perioperative Optimization of Senior Health (POSH) clinic
  Interventions: Other: Process Mapping: Observations; Other: Process Mapping: Interviews; Other: Process Mapping: Focus Group; Other: Participatory Design

INTERVENTIONS:
Other: Process Mapping: Observations — Direct observations of the POSH clinic visit.
Other: Process Mapping: Interviews — Semi-structured interviews of patients and providers involved in the POSH clinic.
Other: Process Mapping: Focus Group — Focus group of providers and staff who conduct the POSH clinic.
  Groups: Healthcare providers
Other: Participatory Design — Participatory design, also called "co-design" is a systems engineering approach where the researchers and participants work together in designing the workflow of an intervention. There will be two groups (design teams) of patients/caregivers and healthcare professionals per location, for a total of four groups.

SUMMARY:
The researchers will conduct observations, interviews, and focus groups with clinicians, staff and patients of the Perioperative Optimization of Senior Health (POSH) clinic, which conducts preoperative comprehensive geriatric assessments (pCGA) at UW Health to understand clinic processes and potential areas for improvement. The goal is to (1) create a process map describing clinic workflow and (2) redesign the process with healthcare providers and patients/families.

DETAILED DESCRIPTION:
Aim 1: Process mapping using direct observation, interviews and focus groups to identify opportunities for system redesign

The research team will directly observe n=30 patients in POSH clinic visits, taking notes and documenting the persons, tasks, tools/technologies, environment and organizational factors affecting healthcare delivery. Observer notes will be supplemented with audio recording of the clinic visit. Observations will also include assessments performed by social workers, pharmacist, medical assistants.

Semi-structured qualitative interviews with patients who participated in the observations and their caregivers, if any, will be conducted 2 weeks after the pCGA visit. Interviewers will assess barriers, facilitators, motivation, and adherence to tasks, and reflections on the process of scheduling, attending and participating in the clinic. Surgeons who refer patients (n=20) will be interviewed using semi-structured guides to elicit feedback on the process map and explore perceived barriers and facilitators to adoption of the pCGA.

Focus Groups: Healthcare professionals and staff (n=20) who conduct the pcga will participate in a focus group to provide feedback on the process map. The researchers will elicit feedback on the process map, clarifying its accuracy as a representation of the tasks and procedures performed, and identifying system-level barriers and facilitators at each step.

Aim 2: Co-design an implementation package for the pCGA at (2a) a large academic hospital and (2b) an affiliate community site.

The research team will apply user-centered participatory design methods to adapt the process map (aim 1) into an implementation package, which consists of a set of implementation strategies, to address barriers and enhance facilitators at each step. Participatory design (also called "co-design") is a systems engineering approach where the researchers and participants work together in designing the workflow of an intervention. Co-design sessions will be conducted in parallel at our University Hospital (2a) and a local affiliated community hospital (2b). There will be two groups (design teams) of patients/caregivers and healthcare professionals per location, for a total of four groups.

This study will include five co-design videoconference sessions with up to n=10 members in each group (total n=40) over approximately 6 months, with 2-3 weeks between each session. Each session will last 90 minutes. The sessions will identify process changes that can address barriers and facilitators to promote implementation of the pCGA. The research team will analyze audio recordings and notes from each session. These findings will be synthesized and presented at the next design session. Each design team will participate in sessions independently, however, the research team will summarize output from each session and provide this content to the alternate design team for comment.

Design sessions are expected to generate an implementation package that is ready for feasibility and pilot testing at the University hospital. Design sessions at the community site will serve as a template for implementation at a future date.

ELIGIBILITY:
Inclusion Criteria:

* Being a patient seen for a pCGA clinic at the time of observations, or being the caregiver of such a patient.
* Being a clinician or staff member working at the pCGA clinic
* Being a surgeon who frequently refers patients to the pCGA clinic

Exclusion Criteria:

* For patients:

  * not being fluent in English
  * having an enacted power of attorney indicating that the patient is unable to make medical decisions for themselves and a legally authorized representative (LAR) does not attend the pCGA visit with the patient
* For pCGA clinicians and staff: none
* For surgeons: none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Observations and Interviews in the Perioperative Optimization of Senior Health (POSH) clinic.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Process map | 12 months
  The direct observations, interviews and focus groups conducted with patients and caregivers will help create a detailed process map of preoperative geriatric assessments. Specifically this map will detail the persons, tasks, tools/technologies, environment and organizational factors involved in the process according to the System Engineering Initiative for Patient Safety model.
Implementation Package | 24 months
  Co-design sessions will generate an implementation package, consisting of a set of implementation strategies, that can be piloted for its feasibility and adapted to facilitate preoperative comprehensive geriatric assessment in other settings.

SECONDARY OUTCOMES:
Qualitative data: Barriers and Facilitators to preoperative comprehensive geriatric assessments | 5 years
  The qualitative analysis performed of interviews and focus groups during process mapping will identify barriers and facilitators to the use of preoperative comprehensive geriatric assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Julia R Berian, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Implementation Pilot of Preoperative CGA Before Major Surgery — https://clinicaltrials.gov/study/NCT06184724